CLINICAL TRIAL: NCT03994055
Title: Effect of an Anti-inflammatory Diet on the Nutritional Status and Cytokine Expression of Patients With Locally Advanced Cervical Cancer: A Randomized Clinical Trial
Brief Title: Effect of an Anti-inflammatory Diet on Patients With Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CEI/1247/17
Record Dates: First submitted 2018-10-18; First posted 2019-06-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer; Uterine Cervical Neoplasm; Pelvic Inflammatory Disease; Radiation Toxicity; Diet Modification
Keywords: Cancer; Intestinal inflammation; Diet
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pelvic Inflammatory Disease; Radiation Injuries; Neoplasms | interventions — Fatty Acids, Omega-3; Antioxidants; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory Diet (Experimental): Dietary intervention providing:
  Energy: 28-31 kcal/kg/day. Protein: 20-30%. Fat: 30-40%. Carbohydrates: 40-50%. The diet will be individualized according to the patients' comorbidities (obesity, type 2 diabetes, hypertension, renal insufficiency).
  This group will include the consumption of foods that contain immune modulating nutrients:
  Omega-3 fatty acids, antioxidants, soluble fiber, probiotics. The recommendation to include these foods will be made according to the patients' access to food in their home area.
  Interventions: Other: Omega-3 fatty acids; Other: Antioxidants; Other: Soluble fiber; Other: Probiotics
- Low residue Diet (Active Comparator): Dietary intervention providing:
  Energy: 28-31 kcal/kg/day. Protein: 20%. Fat: 20%. Carbohydrates: 60%. Diet will have lactose restriction, fiber restriction and fat restriction.
  Interventions: Other: Lactose restriction; Other: Fiber restriction; Other: Fat restriction

INTERVENTIONS:
Other: Omega-3 fatty acids — Diet will include foods rich in omega-3 fatty acids.
  Arms: Anti-inflammatory Diet
Other: Antioxidants — Diet will include foods rich in antioxidant vitamins, trace elements, and polyphenols.
  Arms: Anti-inflammatory Diet
Other: Soluble fiber — Diet will include foods rich in soluble fiber.
  Arms: Anti-inflammatory Diet
Other: Probiotics — Diet will include foods rich in probiotics.
  Arms: Anti-inflammatory Diet
Other: Lactose restriction — Diet will be restricted to 5g lactose/day
  Arms: Low residue Diet
Other: Fiber restriction — Diet will be restricted to 20g fiber/day
  Arms: Low residue Diet
Other: Fat restriction — Diet will be restricted to 20% total energy intake
  Arms: Low residue Diet

SUMMARY:
During radiation therapy (RT) to pelvic tumors, the small intestine, colon and rectum are inevitably included in the radiation field and are healthy tissues that suffer damage as an adverse effect. Pelvic radiation disease (PRD) is the group of gastrointestinal symptoms experienced by patients that receive pelvic radiation. Intestinal inflammation, tissue damage, oxidative stress and tumor metabolism lead the patient to a catabolic state associated with an increase in energy demands. Also, the painful abdominal symptoms restrict the patients' food intake, leading the patients that develop PRD to an increased risk to develop protein-energy malnutrition and micronutrient deficiencies, all of which affect the patients' quality of life. Studies developed in patients with inflammatory bowel disease have suggested that probiotics may have an anti-inflammatory effect in the intestine. In addition, micronutrients and trace elements provide antioxidant capacity and exert immune-modulating effects during periods of intestinal inflammation. Thus, probiotics and immune-modulating nutrients may provide a means to diminish intestinal inflammation and symptoms associated with PRD. In this project the investigators propose that the nutritional management of cervical cancer patients be based on an anti-inflammatory diet, taking into account the nutritional status, age, comorbidities that the patient may present and symptoms developed during treatment. The nutritional intervention will include food rich in immune-modulating nutrients: omega-3 fatty acids, soluble fiber, antioxidants and polyphenols, and probiotics.

DETAILED DESCRIPTION:
Cervical cancer is the second most frequent cancer in Mexican women, representing 16.9% of the total female population. At the National Cancer Institute of Mexico (Instituto Nacional de Cancerología), 80% cervical cancer patients arrive at locally advanced stages (IB2-IVA). Standard treatment for these stages is based on concomitant chemo-radiotherapy. During radiation therapy (RT) to pelvic tumors, the small intestine, colon and rectum are inevitably included in the radiation field and are healthy tissues that suffer damage as an adverse effect. Pelvic radiation disease (PRD) is the group of gastrointestinal symptoms experienced by patients that receive pelvic radiation. Acute PRD occurs during the time of treatment in 60 to 80% patients, symptoms include nausea, diarrhea, tenesmus, abdominal pain, urgency, mucositis, anorexia, bleeding and fatigue; these symptoms limit cancer treatment and affect the patients' quality of life. Chronic PRD is a progressive condition and a problem for cervical cancer survivors, symptoms include altered intestinal traffic, altered intestinal motility and nutrient malabsorption. The intestinal immune system plays an important role in the development of PRD and the secondary effects of RT. Intestinal inflammation, tissue damage, oxidative stress and tumor metabolism lead the patient to a catabolic state associated with an increase in energy demands. Also, the painful abdominal symptoms restrict the patients' food intake, leading the patients that develop PRD to an increased risk to develop protein-energy malnutrition and micronutrient deficiencies, all of which affect the patients' quality of life. Among some of the nutritional intervention assays for patients with PRD, some have described that a low residue diet, restricted in fat (20-25%), lactose (5g) and fiber (20g), reduces the frequency and severity of diarrhea; however, this dietary intervention does not prevent weight loss or malnutrition in patients. Furthermore, low residue diets limit the beneficial effect of dietary fiber and fatty acids that may aid in the inflammatory response. Likewise, patients with inflammatory bowel disease (IBD) develop similar symptoms to PRD. Studies developed in these patients have suggested that probiotics may have an anti-inflammatory effect in the intestine. In addition, micronutrients and trace elements provide antioxidant capacity and exert immune-modulating effects during periods of intestinal inflammation. Thus, probiotics and immune-modulating nutrients may provide a means to diminish intestinal inflammation and symptoms associated with PRD. In this project the investigators propose that the nutritional management of cervical cancer patients be based on an anti-inflammatory diet, taking into account the nutritional status, age, comorbidities that the patient may present and symptoms developed during treatment. The individualized energy requirements and nutrient proportions for patients without comorbidities, and for patients with comorbidities such as obesity, type 2 diabetes, hypertension and renal dysfunction, will be calculated according to the recommendations derived from the Consensus of Nutrition in patients with cancer treated with chemo-radiotherapy to the abdominopelvic area. Furthermore, the nutritional intervention will include food rich in immune-modulating nutrients: omega-3 fatty acids, soluble fiber, antioxidants and polyphenols, and probiotics. Because the low residue diet is routinely used for patients that receive pelvic radiation in other institutions, the anti-inflammatory nutritional intervention will be compared with the low residue diet.

An open controlled randomized clinical trial will be performed on women with locally advanced cervical cancer. Candidates will be randomly assigned to one of the two dietary interventions. Experimental group will receive an anti-inflammatory diet with an energy intake of 28-31 kcal/kg/day, based on 30-40% fat, 20% protein, and 40-50% carbohydrates, the diet will include foods rich in omega-3 fatty acids, soluble fiber, antioxidants and polyphenols, and probiotics. The control group will receive a low residue diet with 28-91 kcal/kg/day, based on 20% fat, 20% protein, and 60% carbohydrates, with no more than 20g fiber and 5g of lactose. In both groups, before, during and after cancer treatment, a thorough nutritional evaluation will be performed, gastrointestinal toxicity will be assessed, and serum cytokine levels and fecal calprotectin and lactoferrin levels will be determined to establish the local and systemic inflammatory response. The quality of life of patients will also be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the study and provide informed consent.
* ECOG: 0-2.
* Willingness to assist to every programed visit, to keep to the dietary intervention and lab tests.
* Diagnosed with cervical cancer.
* Clinical stages IB-2-IVA.
* Candidate to receive concomitant chemo-radiotherapy followed by brachytherapy.
* Disease measured by CT scan.
* No previous treatment based on chemo-radiotherapy. Hemoglobina levels >10g/dL.
* Leucocytes >4000/mm3.
* Platelets > 100000/mm3.
* Adequate hepatic function.

Exclusion Criteria:

* Patients under nutritional treatment or supplement.
* Patients with active uncontrolled infections.
* Patients under treatment with an experimental drug.
* Patients with fistula at the moment of diagnosis.
* Patients with previous malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation, 6 months after treatment initiation
  weight/height squared
Change in levels of IFN-g [pg/ml] | Baseline, 3 weeks after treatment initiation, 6 months after treatment initiation
  Determination of serum IFN-g using immune assay ELISA
Change in levels of calprotectin [pg/ml] | Baseline, 3 weeks after treatment initiation, 6 months after treatment initiation
  Measurement of fecal calprotectin using immune assay ELISA

SECONDARY OUTCOMES:
Change in Gastrointestinal toxicity symptoms grading (severity) scale using the Common Toxicity Criteria for Adverse Events (CTCAE v4) | Baseline, 3 weeks, 12 weeks, 6 months
  Evaluation of the severity of gastrointestinal symptoms according to the Common Toxicity Criteria for Adverse Events (CTCAE v4).
  A grading (severity) scale is provided for each adverse event (AE) term. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4 Life-threatening consequences; urgent intervention indicated.
  Grade 5 Death related to AE.
Change in quality of life summary score using the the quality of life questionnaire specifically developed for cancer patients (EORTC QLQ-C30 v3) | Baseline, 3 weeks after treatment initiation, 12 weeks after treatment initiation, and 6 months after treatment initiation
  Quality of life questionnaire developed and validated for cancer patients (EORTC QLQ-C30 v3, in spanish) will be applied, and the change in summary score will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lucely Cetina, MD, MSc, Study Chair — National Institute of Cancerología
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Shin DW, Nam JH, Kwon YC, Park SY, Bae DS, Park CT, Cho CH, Lee JM, Park SM, Yun YH. Comorbidity in disease-free survivors of cervical cancer compared with the general female population. Oncology. 2008;74(3-4):207-15. doi: 10.1159/000151368. Epub 2008 Aug 20. PMID 18714169
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818
- [Background] Fuccio L, Guido A, Andreyev HJ. Management of intestinal complications in patients with pelvic radiation disease. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1326-1334.e4. doi: 10.1016/j.cgh.2012.07.017. Epub 2012 Jul 31. PMID 22858731
- [Background] Morris KA, Haboubi NY. Pelvic radiation therapy: Between delight and disaster. World J Gastrointest Surg. 2015 Nov 27;7(11):279-88. doi: 10.4240/wjgs.v7.i11.279. PMID 26649150
- [Background] DeWitt T, Hegazi R. Nutrition in pelvic radiation disease and inflammatory bowel disease: similarities and differences. Biomed Res Int. 2014;2014:716579. doi: 10.1155/2014/716579. Epub 2014 May 28. PMID 24982906
- [Background] Wedlake LJ, Shaw C, Whelan K, Andreyev HJ. Systematic review: the efficacy of nutritional interventions to counteract acute gastrointestinal toxicity during therapeutic pelvic radiotherapy. Aliment Pharmacol Ther. 2013 Jun;37(11):1046-56. doi: 10.1111/apt.12316. Epub 2013 Apr 23. PMID 23611411
- [Background] Cetina-Perez L, Castro-Eguiluz D, Onate-Ocana LF. Nutrition in Patients with Cancer Treated with Chemo-radiotherapy to the Abdominopelvic Area. A consensus report. Rev Invest Clin. 2018;70(3):109-111. doi: 10.24875/RIC.18002521. No abstract available. PMID 29943770
- [Background] Castro-Eguiluz D, Leyva-Islas JA, Luvian-Morales J, Martinez-Roque V, Sanchez-Lopez M, Trejo-Duran G, Jimenez-Lima R, Leyva-Rendon FJ. Nutrient Recommendations for Cancer Patients Treated with Pelvic Radiotherapy, with or without Comorbidities. Rev Invest Clin. 2018;70(3):130-135. doi: 10.24875/RIC.18002526. PMID 29943773

DOCUMENTS (1):
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03994055/ICF_000.pdf